CLINICAL TRIAL: NCT04359147
Title: The Role of Stress Neuromodulators in Decision Making Under Risk
Brief Title: The Role of Stress Neuromodulators in Decision Making Under Risk and Selective Attention to Threat
Acronym: SID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katja Wingenfeld, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: WI-3396-3
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Yohimbine; Hydrocortisone; Yohimbine + Hydrocortisone; Placebo
MeSH Terms: interventions — Yohimbine; Administration, Oral; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Yohimbine (Active Comparator): 10 mg
  Interventions: Drug: "Yohimbine"
- Hydrocortisone (Active Comparator): 10 mg
  Interventions: Drug: "Hydrocortisone"
- Yohimbine + Hydrocortisone (Active Comparator): 10 mg each
  Interventions: Drug: "Yohimbine + Hydrocortisone"
- Placebo (Placebo Comparator)
  Interventions: Drug: "Placebo"

INTERVENTIONS:
Drug: "Yohimbine" — Effects on neural correlates of decision-making under risk and selective attention to threat
  Other Names: Pill (oral administration)
  Arms: Yohimbine
Drug: "Hydrocortisone" — Effects on neural correlates of decision-making under risk and selective attention to threat
  Other Names: Pill (oral administration)
  Arms: Hydrocortisone
Drug: "Yohimbine + Hydrocortisone" — Effects on neural correlates of decision-making under risk and selective attention to threat
  Other Names: Pill (oral administration)
  Arms: Yohimbine + Hydrocortisone
Drug: "Placebo" — Effects on neural correlates of decision-making under risk and selective attention to threat
  Other Names: Pill (oral administration)
  Arms: Placebo

SUMMARY:
Incidental affective states, i.e., affective states can influence decision making and selective attention to threatening information. Acute stress is such an affective state and is a powerful contextual modulator of decision-making processes and selective attention to threat. In terms of physiological and neurohormonal changes, the stress response has been well characterized: Exposure to stress elicits an array of autonomic, endocrine, and behavioral responses. The physiological stress response is mediated by the hypothalamic-pituitary-adrenal (HPA) axis and the locus coeruleus noradrenergic (LC-NA) system with cortisol and norepinephrine (NE) as their end products. There is compelling evidence that the stress hormones cortisol and NE influence cognitive processes. However, only very few studies so far used pharmacological approaches to specify the role of stress neuromodulators on decision making and selective attention to threat and these studies are hardly comparable due to differences in the experimental design, e.g., the decision making task used. Furthermore, the neural underpinnings of stress effects on decision making and selective attention to threat are uninvestigated so far. The aim of the proposed project is to clarify the role of the major stress neuromodulators, NE and cortisol, in their contribution to different processes related to decision making under risk and selective attention to threat. To this end, combined precise pharmacological stimulation, behavioral modeling, and fMRI methods will be applied to systematically disentangle the effects of stress hormones on risk attitudes and loss aversion as well as their relation to neural correlates of processing subjective value and risk. Using pharmacological manipulation, the influence of noradrenergic and glucocorticoid activity on decision making under risk at the behavioral, computational, and neural level will be investigated. In addition, the influence of noradrenergic and glucocorticoid activity on selective attention to threat at the behavioural and neural level using a dot-probe paradigm with fearful and neutral faces will be examined. Participants are randomly assigned to one of four groups: (A) yohimbine, (B) hydrocortisone, (C) yohimbine and hydrocortisone, or (D) placebo.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* High-school diploma

Exclusion Criteria:

* Former and present DSM-5 axis I disorders according to the Structured Clinical Interview for DSM (SCID)
* Permanent medication of any kind
* Medical conditions associated with adrenal dysfunction or well-known impact on HPA activity or cognitive function
* Steroid use

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Risk and loss-aversion, choice consistency | 45 minutes
  Behavioural outcome of the decision-making under risk task modeled using prospect theory (PT)
Patch-leaving times | 45 minutes
  Behavioural outcome of the decision-making under risk task including a foraging task part using marginal value theory
Attentional bias to fearful faces | 12 minutes
  Behavioural outcome of the dot-probe task
Blood-oxygen-level-dependent (BOLD) response | 45 + 12 minutes
  In both tasks

SECONDARY OUTCOMES:
Salivary cortisol | 3 hours
  Treatment check
Salivary alpha amylase | 3 hours
  Treatment check
Systolic and diastolic blood pressure | 3 hours
  Treatment check
Heart rate | 3 hours
  Treatment check

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rosada C, Lipka R, Metz S, Otte C, Heekeren H, Wingenfeld K. Effects of stress-related neuromodulators on amygdala and hippocampus resting state functional connectivity. J Psychopharmacol. 2024 Jul;38(7):604-614. doi: 10.1177/02698811241260972. Epub 2024 Jun 20. PMID 38902928